CLINICAL TRIAL: NCT03565354
Title: Efficacy of Preoperative Intravenous Iron Isomaltoside in Colorectal Cancer Surgical Patients With Iron Deficiency Anaemia Compared to Standard Care: a Pilot Randomized Controlled Trial
Brief Title: Efficacy of Preoperative Intravenous Iron in Anaemic Colorectal Cancer Surgical Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Prince of Wales Hospital, Shatin, Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Pui Lam Polly FUNG, Resident trainee, Prince of Wales Hospital, Shatin, Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NTEC-2018-0169
Record Dates: First submitted 2018-05-28; First posted 2018-06-21 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Anemia, Iron-Deficiency; Colorectal Cancer
Keywords: Patient blood management
MeSH Terms: conditions — Anemia, Iron-Deficiency; Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment arm (Active Comparator): intravenous iron isomaltose 3-10 weeks before operation date. The dose will be determined by the patient's body weight: > 50kg: 1000mg; <50kg: 20mg/kg body weight, to be infused over 30 minutes. 2 weeks after intravenous iron isomaltoside administration, blood test for hemoglobin level and iron profile would be repeated. Subjects with hemoglobin level less than 10g/dL will receive a second dose of intravenous iron isomaltoside. The second dose would be identical to the first dose
  Interventions: Drug: iron isomaltoside(Monofer®)
- Control arm (No Intervention): Patient randomized to the control arm will follow the standard perioperative care and the perioperative management they received will be identical to the treatment arm except no intravenous iron isomaltoside will be given.

INTERVENTIONS:
Drug: iron isomaltoside(Monofer®) — intravenous iron isomaltoside
  Arms: Treatment arm

SUMMARY:
Iron deficiency anaemia is a common condition among colorectal surgical patient. Untreated anaemia would lead to increase in blood transfusion, surgical complications and mortality. Treatment with oral iron sulphate is poorly tolerated due to side effects. Intravenous iron supplement provides an alternative way to rapidly replace iron deficit during the preoperative period among surgical patients. Evidence is growing for its effect in rising hemoglobin level and reducing blood transfusion, at the same time supporting its safety profile.

The investigators plan for a single-centered, randomized controlled trial to examine the effect of intravenous iron compared to standard care in terms of hemoglobin level/serum ferritin increment, need for blood transfusion, duration of hospital stay, quality of recovery and surgical complication rate, as well as safety profile among colorectal cancer surgical patients in Hong Kong. The investigator propose the following pilot RCT for exploring the effect size and study process in conducting the above-mentioned large-scale RCT.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years old with written informed consent
* Anaemia defined as: hemoglobin concentration < 13g/dL (same cut-off for both male and female patients according to the International consensus statement on the perioperative management of anaemia and iron deﬁciency)2
* Laboratory test confirmed iron deficiency: serum ferritin <30mcg/L alone or serum ferritin 30-100mcg/L with TSAT < 20%

Exclusion Criteria:

* Pregnancy or lactation
* Other known causes of anaemia apart from iron deficiency: untreated B12/folate deficiency, hemolytic disease, hemoglobinopathy/thalassemia, chronic renal failure on dialysis
* Presence of iron overload (serum ferritin > 300g/dL or TSAT > 50%); known hemochromatosis
* Previous or ongoing iron replacement/use of erythropoietin within 12 weeks before recruitment
* Known hypersensitivity towards iron isomaltoside
* Significant liver function derangement (AST/ALP exceeding three times upper limit of normal range)
* Participation in another ongoing interventional clinical trial(s)
* Patients with less than 3 weeks waiting time to surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Preoperative change in hemoglobin concentration (g/dL) | 3 weeks to 10 weeks
  the difference between the value at diagnosis(baseline) and preoperative day (3-10weeks after diagnosis).
Preoperative change in serum ferritin (mcg/L) | 3 weeks to 10 weeks
  the difference between the value at diagnosis(baseline) and preoperative day (3-10weeks after diagnosis).

SECONDARY OUTCOMES:
Units of red blood cells transfused in perioperative period | 3 weeks to 12 weeks
  Units of red blood cells transfused from diagnosis to discharge
Duration of hospital stay (days) | 1 days up to 1 month
Quality of recovery as measured by questionnaire (QoR-15(Chinese)) | post op day 3
Incidence of adverse reactions/serious adverse events to intravenous iron administration and adverse reaction to blood transfusions | up to post op day 30
Rate of surgical complications | up to post op day 30
  recorded and graded according to Clavien Classification of Surgical Complications
Days (alive and) at home within 30 days of surgery (DAH30) | up to post op day 30

OTHER OUTCOMES:
Patient recruitment rate(%) | through study completion, an average of 1 year
  number of recruited patients divided by number of eligible patients x 100%
Number of patients recruited per month | through study completion, an average of 1 year
Median waiting time to surgery (days) | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fung PLP, Lau VNM, Ng FF, Leung WW, Mak TWC, Lee A. Perioperative changes in haemoglobin and ferritin concentrations from preoperative intravenous iron isomaltoside for iron deficiency anaemia in patients with colorectal cancer: A pilot randomised controlled trial. PLoS One. 2022 Jun 30;17(6):e0270640. doi: 10.1371/journal.pone.0270640. eCollection 2022. PMID 35771891

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-03): https://cdn.clinicaltrials.gov/large-docs/54/NCT03565354/Prot_SAP_000.pdf